CLINICAL TRIAL: NCT01206179
Title: Effect of Bone Marrow-derived Mesenchymal Stem Cell Transplantation in Reconstructing Human Bone Defects
Brief Title: Treatment of Non Union of Long Bone Fractures by Autologous Mesenchymal Stem Cell
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Royan Institute (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Royan-Bone-004
Record Dates: First submitted 2010-09-20; First posted 2010-09-21 (Estimated); Last update posted 2011-12-14 (Estimated); Status verified 2008-06

CONDITIONS: Nonunion Fractures
Keywords: nonunion fracture bone formation pain relief
MeSH Terms: interventions — Carboxylesterase; Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- non union (Experimental): Patients with nonunion fracture of long bones
  Interventions: Biological: cell injection

INTERVENTIONS:
Biological: cell injection — Injection of mesenchymal cells in fractured zone
  Other Names: Cell transplantation

SUMMARY:
Treatment of nonunion, delayed union and malunion fractures of long bones remains problematic. The definition of nonunion is a failure of the fracture to heal in six months in a patient in whom progressive repair had not been observed radiographically between the third and sixth month after the fracture. First of all good surgical techniques are stable immobilization must be obtained and local sepsis excluded. Then stimulation of the callus is required. Numerous techniques have been developed ranging from invasive interventions (including internal fixation with the use of bone graft or bone graft substitutes) to non invasive procedures (ultrasound and pulsed electromagnetic fields).

Recently, autologous cell therapy was presented as an interesting approach. The concept of such therapies is based on the effect of stem cells presented in the bone marrow and able to be transformed in osteoblast cells. The purpose of this study is to find if mesenchymal stem cells can stimulate bone regeneration in nonunion and delayed union fractures to reduce later surgeries required to augment the healing process and to accelerate the time to healing.

DETAILED DESCRIPTION:
Treatment of nonunion, delayed union and malunion fractures of long bones remains problematic. The definition of nonunion is a failure of the fracture to heal in six months in a patient in whom progressive repair had not been observed radiographically between the third and sixth month after the fracture. Nonunion is a serious complication of a fracture, occurring in 2-10% of patients, as it is associated with high economic and health burden. Many cases are subsequently approached by multiple surgical and nonsurgical modalities. Various devices, under the name of "bone growth stimulators" have been used to enhance healing of the fracture. Recent studies, demonstrated the efficacy of mesenchymal stem cells in regeneration of bone and cartilage tissue. In this study percutaneous injection of mesenchymal stem cells to the site of fracture is performed as an outpatient procedure or during an operative exposure to evaluate its efficacy in enhancing bone regeneration. In the case of small size of bone gap, mesenchymal stem cells are injected into the callus of fracture site through an outpatient procedure under the guide of fluoroscopy. If there is a large bone gap, through a surgical management, mesenchymal stem cells seeded on bone matrix are placed at the site of fracture. Patients are followed by X-Ray examination 1,2,6, and 12 months after treatment.

ELIGIBILITY:
* Inclusion criteria:
* Both genders are eligible
* Nonunion or delayed union diagnosed with X-Ray examination.
* More than 4 cm distance to joint
* Provided written informed consent
* Exclusion criteria:
* Multiple major fracture or untreated major fracture
* Infected fracture
* HIV, hepatitis B or hepatitis C infection at the time of screening
* Pregnant or lactating women
* Diagnosis of cancer
* Active treatment with immunosuppressive drugs or anticoagulant agent
* Known allergic reaction to components of study treatment and/or study injection procedure

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2009-03; Primary Completion 2011-03 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Radiological progression of bone fusion | 3 months
  callus formation in fracture zone

SECONDARY OUTCOMES:
Reduction of pain using VAS | 6 months
  Patients feel less pain during use of fractured limb
Cost analysis based on length of hospital stay | 6 months
  Cost benefit of cell transplantation by reduction of hospital admission time

CONTACTS AND LOCATIONS:
Overall Officials: Hamid Gourabi, PhD, Study Chair — President of Royan Institute; Mohammad reza Baghban Eslami Nejad, PhD, Study Director — Sientific Board; Mohssen Emadeddin, MD, Principal Investigator — Orthopadic Investigator; Nasser Aghdami, MD,PhD, Principal Investigator — Head of Regenerative center; Ahmad Vosough, MD, Principal Investigator — Radiologist investigator
Locations (1):
- Royan Institute, Tehran, Iran

REFERENCES:
- [Derived] Emadedin M, Labibzadeh N, Fazeli R, Mohseni F, Hosseini SE, Moghadasali R, Mardpour S, Azimian V, Goodarzi A, Ghorbani Liastani M, Mirazimi Bafghi A, Baghaban Eslaminejad M, Aghdami N. Percutaneous Autologous Bone Marrow-Derived Mesenchymal Stromal Cell Implantation Is Safe for Reconstruction of Human Lower Limb Long Bone Atrophic Nonunion. Cell J. 2017 Apr-Jun;19(1):159-165. doi: 10.22074/cellj.2016.4866. Epub 2016 Dec 21. PMID 28367426
- [Derived] Labibzadeh N, Emadedin M, Fazeli R, Mohseni F, Hosseini SE, Moghadasali R, Mardpour S, Azimian V, Ghorbani Liastani M, Mirazimi Bafghi A, Baghaban Eslaminejad M, Aghdami N. Mesenchymal Stromal Cells Implantation in Combination with Platelet Lysate Product Is Safe for Reconstruction of Human Long Bone Nonunion. Cell J. 2016 Fall;18(3):302-309. doi: 10.22074/cellj.2016.4557. Epub 2016 Aug 24. PMID 27602311
- See also: Related Info — http://www.royaninstitute.org